CLINICAL TRIAL: NCT06143826
Title: Progressive Muscle Relaxation Exercise on Care Burden, Depression, Anxiety and Stress Levels in Dementia Caregivers
Brief Title: Progressive Muscle Relaxation Exercise on Care Burden, Depression, Anxiety, and Stress Levels in Dementia Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Dilek Baykal, Assistant Professor, Atlas University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24246
Record Dates: First submitted 2023-11-11; First posted 2023-11-22 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Caregiver Burden; Dementia
MeSH Terms: conditions — Caregiver Burden; Dementia

STUDY DESIGN:
Intervention Model Description: The research is a pre-test, post-test, cross-sectional, descriptive research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dementia caregiver (Experimental): Caregivers will be asked to perform progressive muscle relaxation exercises 3 days a week for 3 months.
  Interventions: Other: Progressive muscle relaxation exercises

INTERVENTIONS:
Other: Progressive muscle relaxation exercises — Progressive muscle relaxation exercises involve contracting and relaxing 16 muscle groups in the body (hand, upper arm, forearm, forehead, nose, cheek, chin, neck, shoulder, chest, abdomen, waist, stomach, calf, hip, foot). During the exercise, the individual perceives the changes in the muscles during the contraction and relaxation of the muscles. Relaxation exercise is applied along with correct and deep breathing.

SUMMARY:
Dementia, which leads to deterioration in cognitive and behavioral functions, is a chronic progressive disease. Since the diagnosis is made, the care needs of the patients increase. In the later stages of the disease, it becomes completely dependent on the caregiver.

they are coming. Caregiving is performed by family members in developing countries such as Turkey. Family members face many difficulties in their social, work, and daily lives after they start to care. These difficulties are the burden of caregiving is called. Caregivers who perceive the burden of care also experience anxiety, stress, and depression. Jacobson progressive muscle relaxation in coping with these problems exercises can be used. This study was planned to examine the effects of progressive muscle relaxation exercises on anxiety, stress, depression, and caregiver burden in dementia caregivers.

DETAILED DESCRIPTION:
The research is a pre-test, post-test, and cross-sectional research. After explaining the purpose of the study to the caregivers who met the inclusion criteria, the Information Form, the Depression Anxiety Stress-21 Scale (DAS-21), and the Zarit Care Burden Scale will be administered. Then, progressive muscle relaxation exercises will be applied to caregivers. During the interview, the audio recording of the exercise will be given to them. Also, contact information (caregiver and researcher) will be shared mutually.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old
* Being literate
* Not having difficulties in verbal communication
* Have been caring for at least 3 months
* Being able to provide care for free
* Being the primary caregiver of the patient
* Not having a psychiatric diagnosis
* Not using medication for psychiatric illness

Exclusion Criteria:

* Providing care for less than 3 months
* Providing paid care

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Caregiver burden | At the end of the 3 months, the Zarit caregiver burden scale will be applied.
  The Zarit caregiver burden scale will be evaluated before and after the intervention. Five-point Likert-type scale and it consists of 22 statements. The scale has no subgroups. According to the score obtained from the scale: 88-61 points is a severe burden, 60-41 points is moderately severe, 40-21 points is mild to moderate, and less than 21 points is a mild or no burden.

SECONDARY OUTCOMES:
Depression, anxiety and stress | At the end of the 3 months, the Depression, anxiety and stress scale-21 will be applied.
  Depression, anxiety and stress scale will be evaluated before and after the intervention. There are 7 items each to measure depression, anxiety, and stress dimensions on the scale. The first 7 questions in the scale are anxiety, the 7 questions between 8-14 are depression, and last 7 questions 15-21 are also about stress. It is a 4-point Likert type. High scores from the scale indicate depression, anxiety and stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Alzheimer daily life home, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided